CLINICAL TRIAL: NCT04892264
Title: Randomized Phase 1 / 2 Trial of Belantamab Mafodotin, Lenalidomide, and Daratumumab in Relapsed or Newly Diagnosed Multiple Myeloma Patients
Brief Title: Belantamab Mafodotin, Lenalidomide, and Daratumumab for the Treatment of Relapsed, Refractory, or Previously Untreated Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low/slow accrual - did not proceed to Phase 2
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1989; NCI-2021-03479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-009533 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Plasma Cell Myeloma; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (belantamab mafodotin, lenalidomide, daratumumab) (Experimental): INDUCTION: Patients receive belantamab mafodotin IV over 30 minutes on day 1 of odd number cycles, lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Beginning cycle 13, patients receive belantamab mafodotin IV over 30 minutes on day 1 of odd number cycles (starting cycle 13), lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on day 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Belantamab Mafodotin; Biological: Daratumumab; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Procedure: Biospecimen Collection; Procedure: Skeletal Survey X-Ray; Procedure: Low Dose Computed Tomography of the Whole Body; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy
- Arm B (belantamab mafodotin, lenalidomide, daratumumab, Dxevo) (Experimental): INDUCTION: Patients receive belantamab mafodotin IV over 30 minutes on day 1 of cycles 2, 4, 6, 8, 10, and 12, lenalidomide PO QD on days 1-21, daratumumab IV over 90 minutes on days 1, 8, 15, and 22 of cycles 1 and 3, and days 1 and 15 on cycles 5, 7, 9, and 11. Patients also receive dexamethasone PO on days 1, 8, 15 and 22. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Beginning cycle 13, patients receive belantamab mafodotin IV over 30 minutes on day 1 of even numbered cycles, lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on day 1 of odd numbered cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Belantamab Mafodotin; Biological: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Procedure: Biospecimen Collection; Procedure: Skeletal Survey X-Ray; Procedure: Low Dose Computed Tomography of the Whole Body; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Biological: Belantamab Mafodotin — Given IV
  Other Names: Belantamab Mafodotin-blmf; Blenrep; GSK2857916; J6M0-mcMMAF
Biological: Daratumumab — Given IV
  Other Names: Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm B (belantamab mafodotin, lenalidomide, daratumumab, Dxevo)
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Skeletal Survey X-Ray — Undergo X-ray skeletal survey
  Other Names: Skeletal Survey
Procedure: Low Dose Computed Tomography of the Whole Body — Undergo whole body low dose CT
  Other Names: Low-dose Whole-body CT; Whole Body Low Dose Computed Tomography; Whole Body Low Dose CT; Whole-body Low-dose CT
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow

SUMMARY:
This phase I/II trial studies the best dose and effect of belantamab mafodotin given together with lenalidomide and daratumumab in treating patients with multiple myeloma that has come back (relapsed), does not respond to treatment (refractory) or for which the patient has not received treatment in the past (previously untreated). Belantamab mafodotin is a monoclonal antibody, called belantamab, linked to a chemotherapy drug, called mafodotin. Belantamab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as BCMA receptors, and delivers mafodotin to kill them. Lenalidomide is an immunomodulatory drug (altering the immune effects on the tumor cell). Daratumumab is a drug that is a monoclonal antibody that is directed towards a protein on the myeloma cell. Giving belantamab mafodotin together with lenalidomide and daratumumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of belantamab mafodotin (belantamab) in combination with daratumumab and lenalidomide in patients with relapsed or refractory multiple myeloma. (Phase I) II. To assess the confirmed complete response rate following induction therapy with belantamab, daratumumab, and lenalidomide (bortezomib-dexamethasone-rituximab [BDR]), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone, when used as initial therapy in patients with previously untreated symptomatic multiple myeloma patients. (Phase II)

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with the combination of belantamab, daratumumab, and lenalidomide when used as initial therapy in patients with relapsed multiple myeloma. (Phase I) II. To assess the overall response rate (ORR) and >= very good partial response (VGPR) rate of belantamab, daratumumab, and lenalidomide (BDR) (Phase II), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone. (Phase II) III. To assess the progression free survival and overall survival among patients with previously untreated symptomatic multiple myeloma following treatment with belantamab, daratumumab, and lenalidomide (BDR) (Phase II), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone. (Phase II) IV. To assess the time to response (defined as the time between the date of first dose and the first documented evidence of a partial response or better) following treatment with belantamab, daratumumab, and lenalidomide (BDR) (Phase II), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone. (Phase II) V. To describe the toxicities associated with belantamab, daratumumab, and lenalidomide (BDR) (Phase II), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone. (Phase II)

CORRELATIVE RESEARCH OBJECTIVE:

I. Examine the rate of minimal residual disease (MRD) negativity following induction therapy with the combination of belantamab, daratumumab, and lenalidomide (BDR) (Phase II), OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone. (Phase II)

OUTLINE: This is a phase I dose-escalation study of belantamab mafodotin, followed by a phase II study.

PHASE I:

INDUCTION: Patients receive belantamab mafodotin intravenously (IV) over 30 minutes on day 1, lenalidomide orally (PO) once daily (QD) on days 1-21, and daratumumab IV over 90 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Treatment with belantamab mafodotin repeats every 56 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Treatment with lenalidomide and daratumumab repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning cycle 13, patients receive belantamab mafodotin IV over 30 minutes on day 1 of odd number cycles, lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on day 1. Treatment with belantamab mafodotin repeats every 56 days, and every 28 days for lenalidomide and daratumumab in the absence of disease progression or unacceptable toxicity. Treatment with belantamab mafodotin repeats every 56 days (every other cycle) for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Treatment with lenalidomide and daratumumab repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM A:

INDUCTION: Patients receive belantamab mafodotin IV over 30 minutes on day 1 of odd number cycles, lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning cycle 13, patients receive belantamab mafodotin IV over 30 minutes on day 1 of odd number cycles (starting cycle 13), lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on day 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM B:

INDUCTION: Patients receive belantamab mafodotin IV over 30 minutes on day 1 of cycles 2, 4, 6, 8, 10, and 12, lenalidomide PO QD on days 1-21, daratumumab IV over 90 minutes on days 1, 8, 15, and 22 of cycles 1 and 3, and days 1 and 15 on cycles 5, 7, 9, and 11. Patients also receive dexamethasone PO on days 1, 8, 15 and 22. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning cycle 13, patients receive belantamab mafodotin IV over 30 minutes on day 1 of even numbered cycles, lenalidomide PO QD on days 1-21, and daratumumab IV over 90 minutes on day 1 of odd numbered cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo blood sample collection, X-ray skeletal survey or whole body low dose computed tomography (CT), bone marrow aspiration and biopsy throughout study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Phase I: Relapsed or refractory multiple myeloma with at least one prior line of therapy that includes a proteasome inhibitor and an immunomodulatory drug. Patient should be refractory to lenalidomide
* Phase II: Previously untreated multiple myeloma (diagnosed by International Myeloma Working Group [IMWG] criteria) or have received no more than one cycle of Standard of Care treatment regimen
* Note: Prior radiation therapy for the treatment of solitary plasmacytoma is permitted. Prior therapy with clarithromycin, dehydroepiandrosterone (DHEA), anakinra, pamidronate or zoledronic acid is permitted. Any additional agents not listed must be approved by the principal investigator
* Measurable disease

  * Note: Phase I patients can enter trial with M spike >= 0.5 g/dl
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1200/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Prothrombin time (PT)/International Normalized Ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 30 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Female participants: Female participant is eligible to participate if she is not pregnant or breast feeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR
  * Due to lenalidomide being a thalidomide analogue with risk for embryofetal toxicity and prescribed under a pregnancy prevention/controlled distribution program, and bortezomib having the potential to cause fetal harm, WOCBP participants will be eligible if they commit to either:

    * Abstain continuously from heterosexual sexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * To use birth control as follows:

      * Two methods of reliable birth control (one method that is highly effective and one additional effective (barrier) method), beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment. Thereafter, WOCBP participants must use one method of reliable birth control that is highly effective for a further 4 months following discontinuation of belantamab mafodotin or a further 2 months after discontinuation of daratumumab. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of lenalidomide, or 4 months following discontinuation of belantamab mafodotin treatment, whichever is longer.

        * Note: The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy
* Male participants: Male participants are eligible to participate if they agree to the following from the time of first dose of study treatment until 28-days after the last dose of lenalidomide, or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm:

  * Refrain from donating sperm PLUS either
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
  * Must agree to use contraception/barrier as detailed below:

    * Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of < 1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females)
* Ability to understand the study procedures and provide written informed consent
* Negative hepatitis B test (defined by a negative test for hepatitis B surface antigen [HBsAg], or antibodies to hepatitis B surface and/or core antigens [antiHBs or antiHBc])

  * Note: Participants with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior hepatitis B virus (HBV) vaccination do not need to be tested for HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR). Those who are PCR positive will be excluded from the study
* Participant agrees not to use contact lenses while participating in the study
* Willingness to provide mandatory bone marrow and blood specimens for research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* All prior treatment-related toxicities (defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be =< grade 1 at the time of enrolment except for alopecia

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance or smoldering multiple myeloma
* Major surgery =< 28 days prior to registration
* Plasmapheresis =< 14 days prior to registration
* Diagnosed or treated for another malignancy =< 2 years prior to registration or previously diagnosed with another malignancy and have any evidence of residual disease

  * Note: Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
  * Note: If there is a history of prior malignancy, they must not be receiving other specific treatment (hormone therapy, chemotherapy, or immunotherapy) for their cancer
* Receiving any other concurrent chemotherapy, systemic steroids, any ancillary therapy considered investigational for treatment of multiple myeloma, or receiving radiotherapy =< 14 days or five half-lives, whichever is shorter, prior to first dose of study treatment. Note: Bisphosphonates are considered to be supportive care rather than therapy and are thus allowed while on protocol treatment
* Known to be human immunodeficiency virus (HIV) positive
* Presence of positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment

  * Note: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained
  * Note: Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (defined as infection undergoing treatment)
  * Active mucosal or internal bleeding
  * Social situations that would limit compliance with study requirements.
  * Corneal epithelial disease (except for mild changes in the corneal epithelium)
  * Known gastrointestinal disease (including difficulty swallowing) or gastrointestinal procedure that could interfere with the oral absorption or tolerance of lenalidomide or dexamethasone
  * Unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
  * Active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Note: Participants with isolated proteinuria resulting from MM are eligible, provided they fulfill inclusion criteria
* Evidence of cardiovascular disease risk, as defined by any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting =< 90 days prior to registration
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system
  * Uncontrolled hypertension
* History of myocardial infarction, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure) or known sensitivity to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of belantamab in combination with daratumumab and lenalidomide in patients with relapsed and/or refractory multiple myeloma (Phase I) | Up to 28 days
  The MTD will be determined by the dose limiting toxicities (DLTs) seen in cycle 1 of the therapy in the phase I portion. The phase II portion will be based on the determined MTD. MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).
Complete response rate with belantamab, daratumumab, and lenalidomide, OR alternating cycles of daratumumab, lenalidomide, dexamethasone and belantamab, lenalidomide and dexamethasone, when used as initial therapy (Phase II) | After completion of induction therapy
  A confirmed response is defined as a patient who has achieved a stringent complete response (sCR) or CR (as defined by the International Myeloma Working Group criteria) and maintained it on two consecutive evaluations at least 2 weeks apart.

SECONDARY OUTCOMES:
Incidence of toxicity (Phase I) | Up to 3 years
  Defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Overall response rate | Up to 3 years
  Will be estimated by the number of patients with each response category (e.g: sCR, CR, VGPR, partial response [PR], etc) divided by the total number of evaluable patients.
Greater than or equal to very good partial response (VGPR) rate | Up to 3 years
  Will be estimated by the number of patients with each response category (e.g: sCR, CR, VGPR, PR, etc) divided by the total number of evaluable patients.
Progression-free survival | From registration to the earliest date of documentation of disease progression or relapse or death due to any cause, assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier.
Time to response | Time between the date of first dose and the first documented evidence of a partial response or better, assessed up to 3 years
  Descriptive statistics will be estimated.
Incidence of adverse events | Up to 30 days post treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials